CLINICAL TRIAL: NCT02004301
Title: A Pilot Pharmacoscintigraphic Clinical Study to Investigate the Behaviour of Delayed-release Tablets Consisting of a Diclofenac Potassium Core Coated With Barrier Granules, in Healthy Volunteers
Brief Title: A Study to Investigate Delayed-release Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BDD Pharma Ltd (Industry)
Collaborators: Drug Delivery International Ltd (Industry)
Responsible Party: Principal Investigator, Howard Stevens, Chairman, BDD Pharma Ltd
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FM1202A
Record Dates: First submitted 2013-12-02; First posted 2013-12-09 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Pain
Keywords: Formulation behaviour; Drug absorption profile
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiolabelled T4 Tablet (Experimental): Single dose of delayed release diclofenac potassium (25 mg) tablet with time delay of 4 h radiolabelled with 4 MBq 99mTc
  Interventions: Drug: Radiolabelled T4 Tablet
- Radiolabelled T6 Tablet (Experimental): Single dose of delayed release diclofenac potassium (25 mg) tablet with time delay of 6 h radiolabelled with 4 MBq 99mTc
  Interventions: Drug: Radiolabelled T6 Tablet

INTERVENTIONS:
Drug: Radiolabelled T4 Tablet
  Other Names: Delayed release diclofenac potassium tablet
  Arms: Radiolabelled T4 Tablet
Drug: Radiolabelled T6 Tablet
  Other Names: Delayed release diclofenac potassium tablet
  Arms: Radiolabelled T6 Tablet

SUMMARY:
This is a single-centre, open-label, non-randomised, two-arm study in 12 healthy male volunteers. This study is designed to correlate the gastrointestinal transit behaviour of delayed-release diclofenac potassium tablets with their pharmacokinetic (PK) absorption profiles.

We will be looking at:

1. The behaviour of the tablets (when, where and how quickly they break up)
2. The gastric emptying time of the tablets (when they leave the stomach)
3. The gastrointestinal transit of the tablets (how long they take to travel through the gut)
4. Blood levels of the drug (diclofenac)

DETAILED DESCRIPTION:
The tablets being tested will contain the drug, diclofenac potassium. Diclofenac potassium is a non-steroidal anti-inflammatory drug (NSAID) taken to reduce inflammation and as an analgesic, reducing pain in certain conditions such as rheumatoid arthritis, gout and post-operative pain.

The 2 treatments are as follows:

Tablet T4: Radiolabelled delayed release diclofenac potassium tablet with time delay of 4 h

Tablet T6: Radiolabelled delayed release diclofenac potassium tablet with time delay of 6 h

In this study we will be using a type of radioactive material (known as technetium-99m) which is routinely used in investigations of this type. A small amount of technetium-99m will be put into each tablet.

Primary Objective A)To assess the site and time of onset and complete release of radiolabel from two delayed-release diclofenac potassium formulations

Secondary Objectives B)To determine gastrointestinal transit parameters of two delayed-release diclofenac potassium formulations C)To determine the plasma concentrations of diclofenac at each PK sampling point post-administration of two delayed-release diclofenac potassium formulations D)To assess and compare between the two delayed-release diclofenac potassium formulations, as a minimum, the following PK parameters: tlag, tmax, Cmax and AUC0-15h

ELIGIBILITY:
Inclusion Criteria:

- Male 18 to 45 years inclusive. BMI 18.0 to 29.9 kg/m2. Body weight ≥50 kg. Understands and is willing, able and likely to comply with all study procedures and restrictions. Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent.

Good general health with (in the opinion of the Investigator) no clinically significant and relevant abnormalities of medical history or physical examination.

Exclusion Criteria:

Current or recurrent disease that could affect the study conduct or laboratory assessments.

Current or relevant previous history of serious, severe or unstable physical or psychiatric illness, any medical disorder that may require treatment or make the subject unlikely to fully complete the study, or any condition that presents undue risk from the study medication or procedures.

History of current or relevant previous non self-limiting gastrointestinal disorders, in particular, peptic ulcer disease and/or gastrointestinal bleeding.

History of hypersensitivity to aspirin or any other NSAID. Currently suffering from disease known to impact gastric emptying, e.g. migraine, insulin-dependent diabetes mellitus.

Laboratory screening results that suggest an abnormal liver and/or renal function.

Subject has a screening QTc value of greater than or equal to 450 msec or an ECG that is not suitable for QTc measurements.

The physician responsible considers the volunteer unfit for the study. Taken prescribed medication within 14 days prior to the first Assessment Visit which, in the opinion of the physician responsible, will interfere with the study procedures or compromise safety.

Taken over-the-counter (OTC) medication within 48 hours prior to the first Assessment Visit. Subjects may still be entered into the study if, in the opinion of the physician responsible, the medication will not interfere with the study procedures or compromise safety. The occasional use of paracetamol for pain relief (within its labelled dosage) is permitted but must not be taken within 48 hours of an Assessment Visit.

Recent history (within the last year) of alcohol or other substance abuse. Average weekly alcohol intake of greater than 21 units. Positive urine drugs of abuse test at screening. Note: At the discretion of the Investigator, the test may be repeated Positive breath alcohol test at screening. Recently discontinued smoking (less than 3 months). Currently a smoker or user of nicotine-containing products. Allergy to a drug, to any component of the dosage form or any other allergy. Vegetarian. Lactose intolerant. Allergy to any of the contents of the standard dinner.

Participation in another clinical study (inclusive of final post-study examination) or receipt of an investigational drug within the 12 weeks before first screening visit.

Previous participation in this study. Will result in a participation in more than four studies over a twelve month period.

An employee of the sponsor, client or study site or members of their immediate family.

Will exceed the limits of total radiation exposure allowed in any 12 month period (5 mSv), or will exceed 10 mSv over any three year period.

Intending to father a child in the 3 months following the study or are unwilling to abstain from sexual intercourse with pregnant or lactating women Unwilling to use a condom/spermicide in addition to having their female partner use another form of contraception such as an IUD, diaphragm with spermicide, oral contraceptives, injectable progesterone, subdermal implants or a tubal ligation if the woman could become pregnant from the time of the first Assessment Visit until 3 months following the study.

Donated blood or experienced significant blood loss within 3 months of screening and for the duration of the study.

Difficulty in accessibility of forearm veins. Any non-removable metal objects in their chest or abdominal.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Scintigraphic analysis of time and site of onset and complete release of radiolabel | 15 hours

SECONDARY OUTCOMES:
Pharmacokinetic (PK) absorption profiles and parameters of diclofenac | 15 hours

CONTACTS AND LOCATIONS:
Overall Officials: Howard NE Stevens, PhD, Principal Investigator — BDD Pharma Ltd
Locations (1):
- Bio-Imaging Centre, Basement Medical Block, Within Glasgow Royal Infirmary, 84 Castle Street, Glasgow, United Kingdom